CLINICAL TRIAL: NCT06472388
Title: Randomized Phase II Trial of Everolimus 5 mg vs 10 mg/Daily for Patients With Advanced Neuroendocrine Tumors
Brief Title: Everolimus 5 mg vs 10 mg/Daily for Patients With Neuroendocrine Tumors
Acronym: EVENET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Riechelmann, Dr, AC Camargo Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67420523.4.1001.5432
Record Dates: First submitted 2024-05-03; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Neuroendocrine Tumors; Progression; Neuroendocrine Tumor Grade 1; Neuroendocrine Tumor Grade 2; Neuroendocrine Tumor of Pancreas; Neuroendocrine Tumor of the Lung; Neuroendocrine Tumor Carcinoid
MeSH Terms: conditions — Neuroendocrine Tumors; Disease Progression; Adenoma, Islet Cell; Carcinoid Tumor | interventions — Everolimus

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, phase II near-equivalence clinical trial of oral everolimus 5 mg vs 10 mg oral/daily and continuously in patients with Grade 1 or Grade 2 metastatic NET, with tumor progression or intolerance to at least one line of treatment and with radiological disease progression within 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Everolimus 5 (Experimental): oral everolimus 5 mg/daily continuously until progression or intolerance or consent withdrawal. dose reduction for toxicity is allowed.
  Interventions: Drug: Everolimus 5 MG
- Everolimus 10 (Active Comparator): oral everolimus 10 mg/daily continuously until progression or intolerance or consent withdrawal. dose reduction for toxicity is allowed.
  Interventions: Drug: Everolimus 5 MG

INTERVENTIONS:
Drug: Everolimus 5 MG — oral everolimus 5 mg/daily

SUMMARY:
Everolimus is approved in many countries to treat patients with advanced/metastatic well-differentiated neuroendocrine tumors (NET), providing median progression-free survival times of approximately 12 months across different types of NET. However, it is can cause severe adverse effects. Phase I trial demonstrated that a dose of 5mg/day/week was sufficient to inhibit cell proliferation by blocking the mTOR pathway.

This is a randomized, open-label, phase II near-equivalence clinical trial of oral everolimus 5 mg vs 10 mg oral/daily and continuously in patients with Grade 1 or Grade 2 metastatic NET, with tumor progression or intolerance to at least one line of treatment and with radiological disease progression within 6 months.

DETAILED DESCRIPTION:
Everolimus toxicity can also be serious, requiring hospital medical assistance. In a study with more than 100 Latin American patients led by our group, approximately 20% of patients with NET treated with everolimus 10mg/day had serious infections, such as pneumonia, abscesses, pyelonephritis, with 7% developing opportunistic infections, such as toxoplasmosis and pneumocystosis, requiring hospital admissions.

The rationale for testing 5mg/day comes from the results of phase I trials of everolimus, where a dose of 5mg/day was sufficient to inhibit cell proliferation by blocking the mTOR pathway.

Therefore, everolimus 5mg/day appears to have antitumor effects equivalent to 10mg/day, but it is less toxic than 10mg/day. Retrospective data from our center also suggest that 5mg is similar to 10mg/daily in terms of time to treatment failure in patients with advanced NETs (unpublished data).

Objectives:

* To evaluate whether everolimus at a dose of 5 mg/day may be as effective, but safer, as 10 mg/day in the treatment of patients with advanced NET.
* To compare progression-free survival and time to treatment failure between study arms
* To compare radiological response using RECIST v.1.1 criteria.
* To compare the frequency of grade > 1 toxicities using CTCAE v.5.0.
* To assess tolerability by measuring the frequency and intensity of adverse events measured by the CTCAE version 5.0 criteria and the need for temporary or permanent interruption of everolimus.

Methods:

Randomized, open-label, phase II near-equivalence clinical trial of oral everolimus 5 mg vs 10 mg oral/daily and continuously in patients with Grade 1 or Grade 2 metastatic NET, with tumor progression or intolerance to at least one line of treatment and with radiological disease progression within 6 months.

Eligibility criteria:

Inclusion:

* Histological confirmation of well-differentiated Grade 1/Grade 2 NET from gastrointestinal, pancreatic, pulmonary or unknown primary sites.
* Metastatic or locally advanced and unresectable disease, measurable by images
* Disease progression by RECIST 1.1 in the last 6 months assessed by local investigators
* At least one previous line of systemic treatment (suspended for more than 3 weeks).
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Good organ function:

  * Hemoglobin > 8 g/dL
  * Neutrophils ≥ 1,500/mm³
  * Platelets > 90,000/mm³
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN [upper limit of normal] or ≤ 5 x ULN for patients with liver metastases
  * Bilirubin ≤ 1.5 x ULN, creatinine < 1.5 mg/dL

Concomitant use of somatostatin analogues is allowed for patients with functioning NET.

Exclusion:

* Aggressive disease requiring cytotoxic therapy
* Severe/uncontrolled comorbid conditions that deem participant unfit for everolimus therapy, as per investigators' judgement.
* MiNEN

Procedures:

Randomization 1:1 will be performed centrally by RedCap software at AC Camargo Cancer Center, Sao Paulo, Brasil.

* Group 5 mg: participants will receive everolimus at a dose of 5 mg, orally, per day, continuously
* Group 10 mg group: participants will receive everolimus at a dose of 10 mg, orally, per day, continuously

The participant will receive everolimus 5mg or 10mg and must take 1 (one) tablet, orally, once a day, after breakfast, starting within 4 weeks from randomization. Every 4 weeks of treatment will correspond to 1 treatment cycle. Before starting each cycle, participants will undergo a medical visit to evaluate undesirable effects, medical history, physical examination and check the results of blood tests.

CT scans (or MRI, if applicable) will be performed at every 3 cycles to assess treatment antitumor effect until progression. The treatment will last until tumor progression by RECIST 1.1, intolerance/ severe adverse effects or consent withdrawal.

Participants will be evaluated clinically and with laboratory tests every 4 weeks until resolution of any adverse effects of the treatment. Patients who receive at least one dose of everolimus will be evaluated for the occurrence of toxicities

Sample size:

N=100 patients (50 per arm)

H0= 50% progression free at 12 months H1= 42% progression free at 12 months (inferior value of the 95% CI, based on RADIANT trials) Alpha error (one-sided) = 5% Beta error = 10% Attrition rate = 20%

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of well-differentiated Grade 1/Grade 2 NET from gastrointestinal, pancreatic, pulmonary or unknown primary sites.
* Metastatic or locally advanced and unresectable disease, measurable by images
* Disease progression by RECIST 1.1 in the last 6 months assessed by local investigators
* At least one previous line of systemic treatment (suspended for more than 3 weeks).
* Eastern Cooperative Oncology Group (ECOG) 0-2 o Good organ function:

  * Hemoglobin > 8 g/dL
  * Neutrophils ≥ 1,500/mm³
  * Platelets > 90,000/mm³
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN [upper limit of normal] or ≤ 5 x ULN for patients with liver metastases
  * Bilirubin ≤ 1.5 x ULN, creatinine < 1.5 mg/dL

Exclusion Criteria:

* Aggressive disease requiring cytotoxic therapy
* Severe/uncontrolled comorbid conditions that deem participant unfit for everolimus therapy, as per investigators' judgement.
* MiNEN

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 12 months | 12 months
  Proportion of patients without radiological progression or death at 12 months from first day of everolimus

SECONDARY OUTCOMES:
progression free survival | 12 months
  Time from first day of everolimus until radiological progression or death (time to event)
time to treatment failure | 12 months
  fTime from first day of everolimus until progression, treatment discontinuation for toxicity or death

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - AC Camargo Cancer Center, São Paulo, São Paulo
  - AC Camargo Cancer Center, São Paulo

IPD SHARING:
Plan to Share IPD: No
No plan yet